CLINICAL TRIAL: NCT00701350
Title: Identification of Proteomic Markers of Intra-amniotic Infection (IAI) in Patients With Preterm Premature Rupture of Amniotic Membranes (PPROM)
Brief Title: Biomarkers of Intra-amniotic Infection in Women With Preterm Premature Ruptured Amniotic Membranes
Acronym: PPROM
Status: Completed | Type: Observational
Sponsor: ProteoGenix, Inc. (Industry)
Collaborators: Obstetrix Medical Group (Industry)
Responsible Party: Durlin Hickok, MD, MPH; Chief Medical Officer, ProteoGenix
Other Study IDs: PGX03-OBX0009
Record Dates: First submitted 2008-06-13; First posted 2008-06-19 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Intra-amniotic Infection; Preterm Birth
Keywords: Pregnancy; Intra-amniotic Infection; Preterm Birth; Preterm Premature Rupture of Membranes
MeSH Terms: conditions — Premature Birth; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cervical-vaginal Fluid, Amniotic Fluid, Maternal Serum, Neonatal Cord Blood, Placental and Umbilical Cord Tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women presenting with preterm gestation and ruptured membranes

SUMMARY:
The purpose of this study is to investigate the expression of protein biomarkers in cervical vaginal fluid in women with preterm premature rupture of membranes (PPROM)

DETAILED DESCRIPTION:
Preterm premature rupture of the membranes (PPROM) prior to 37 weeks of gestation occurs in approximately 3% of all pregnancies and is associated with one-third of all preterm births (Mercer, 2003). While there are multiple possible etiologies of PPROM, intra-amniotic infection has been implicated as a major contributor, especially at early gestational ages where fetal and neonatal adverse sequelae are frequent (Yoon, et al. 2000). Micro-organisms are recovered from the amniotic fluid obtained by trans-abdominal amniocentesis in 25-40% of women at the time of presentation with PPROM (Simhan and Canavan 2005).

Significant risks to the fetus following PPROM include both complications related to prematurity and to infection or inflammation (ACOG Practice Bulletin 2007). Complications related to prematurity include respiratory distress, intraventricular hemorrhage, and necrotizing enterocolitis. IAI, both clinically apparent and occult, is an important and potentially preventable cause of cerebral white matter injury and cerebral palsy. Ideally, an early diagnosis of IAI in the setting of PPROM is important to allow timely treatment and intervention. Amniocentesis is successful from 40 - 72% of the time with PPROM (Garite, 1982, Blackwell and Berry, 1999). Despite the accuracy for determining infection and the feasibility of amniocentesis, the vast majority of clinicians are reluctant and/or unwilling to perform this procedure in this clinical setting (Capeless and Mead, (1987). There is therefore a critical need for a noninvasive test to identify patients with IAI and PPROM. Timely identification of these sub-clinically infected patients is critical in designing rationale and efficacious treatment strategies that may reduce the fetal and neonatal sequelae associated with PPROM.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject has singleton gestation
* Subject has fetus with getstational age of at least 23 0/7 days and no greater than 33 6/7 days
* Subject has diagnosis of preterm premature rupture of amniotic membranes as determined by at least two of the following:

  1. Postive pooling,
  2. Presence of ferning from cervical vaginal fluid swab on an air dried slide,
  3. Postivie nitrizine pH test, or, in lieu of the criteria listed above
  4. Positive Amnisure test result
  5. Positive indigo carmine egress vaginally following instillation at amniocentesis
* Subject is enrolled and has an amniocentesis within 24 hours of membrane rupture
* Subject is a candidate for expectant management as evidenced by the following:

  1. Absence of labor (defined by absence of painful uterine contractions)
  2. No clinical signs of infection (maternal fever of 37.9 C or greater, fetal heart rate greater than 160 bpm, uterine tenderness, purulent aminorrhea)
  3. presence of non-reassuring heart tracing
* Subject is a candidate for amniocentesis as evidenced by the following:

  1. Ultrasound reveals pocket of fluid likely to result in successful amniocentesis
  2. Physician believes that the subject shoudl undergo amniocentesis as part of their routine evaluation of their current problem of PPROM to rule out infection and/or to test for lung maturity

Exclusion Criteria:

* Subject has a fetus with major fetal anomaly (life threatening or requires surgical intervention) or chromosomal aneuploidy
* Subject has pre-existing medical indication for preterm delivery (e.g., pre-eclampsia, refractory hypertension, diabetes with significant complications, active lupus)
* Subject is unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women within the target gestational age range presenting to labor and delivery wards with documented rupture of amniotic membranes no greater than 24 hours duration.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Expression of protein biomarkers in cervial vaginal fluid | 24 hours of amniotic membrane rupture to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Richard Porecco, MD, Principal Investigator — Obstetrix Medical Group
Locations (4):
- United States (4):
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Good Samaritan Hospital, San Jose, California
  - Presbyterian St. Luke's Medical Center, Denver, Colorado